CLINICAL TRIAL: NCT06841068
Title: A Phase I/II Trial of Intrathecal Delivery of Amniotic Fluid Stem Cells for Primary and Secondary Progressive Multiple Sclerosis
Brief Title: Intrathecal Amniotic Fluid Stem Cells for Progressive Multiple Sclerosis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFSC-PMS-001
Record Dates: First submitted 2025-02-16; First posted 2025-02-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis, Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label stem cell arm (Experimental): The first 5 participants will receive 4 intrathecal injections of c-Kit stem cells at a dose of 25 x 106 cells per injection.
  The next 5 patients will receive 4 intrathecal injections of c-Kit stem cells at a dose of 50 x 106cells per injection.
  The next 10 patients will receive 4 intrathecal injections of c-Kit stem cells at a dose of 80 x 106cells per injection.
  Only if a dose is deemed safe by the investigators after 1 month of its first injection, will we advance to the next dose.
  Interventions: Biological: Amniotic fluid or placental CD117 stem cells

INTERVENTIONS:
Biological: Amniotic fluid or placental CD117 stem cells — CD117 (c-Kit) positive stem cells, extracted from ethical fetal sources such as amniotic fluid and placental tissue.

SUMMARY:
In this clinical trial, researchers are exploring a novel approach to delivering therapy directly into the spinal fluid, which surrounds and nourishes the brain and spinal cord. The study focuses on patients with progressive multiple sclerosis (MS), a form of the disease that leads to worsening disability without the typical relapses seen in other MS subtypes.

This investigational therapy involves the use of stem cells derived from amniotic fluid-the protective liquid surrounding a developing baby in the womb. To the best of the researchers' knowledge, these specific stem cells have never been tested in MS patients before. Amniotic fluid is ethically sourced from routine medical procedures during pregnancy, and similar stem cells can also be obtained from placentas that are typically discarded after childbirth.

Participants in the trial will receive multiple injections of these stem cells into their spinal fluid over the course of a year. Researchers will closely monitor for the safety of this therapy, as well as monitor the participants' walking ability and other neurological functions to assess potential improvements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years.
* Diagnosed with primary or secondary progressive MS according to the 2017 revised McDonald criteria.
* Expanded Disability Status Scale (EDSS) of 3.0 to 8.0 with at least one functional scale that is not vision or sensory or brainstem or cognitive or bowel/bladder that is scoring 3.0 or greater.
* Clinically stable as determined by their neurologist for the past 6 months.
* On no disease-modifying therapy (DMT) for at least 6 months, or on the same DMT for at least 6 months before study entry.
* Can give informed consent.
* Women of child-bearing age must practice adequate contraception techniques in the eye of the investigator and continue to do so during the study period.
* Must be a good candidate, known for compliance for example, in the opinion of the investigators.

Exclusion Criteria:

* Participation in another clinical trial within the last 30 days.
* Severe allergic reactions to any component of the study treatments.
* Significant comorbidities.
* Active infections or malignancies.
* History of a malignancy within the past two years except for skin cancer that has been excised and controlled with only surgical treatment, not requiring chemotherapy or radiotherapy.
* Any medical condition that the investigator deems as unsuitable with therapy.
* Prior organ, tissue, or stem cell transplant or cell therapy within 3 years of study entry
* A diagnosis of a progressive neurological disorder other than multiple sclerosis.
* Inability to have an MRI scan.
* Inability to have a lumbar puncture, for example severe bleeding diathesis.
* Pregnant or breastfeeding or intention to become pregnant during the study.
* The results of the following laboratory results deemed suitable by the investigators: CBC with diff, CMP, INR, aPTT, Hepatitis C serology, HIV serology, RPR.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From enrollment to the end of treatment at 12 months
  The primary safety outcome will be the incidence of adverse events (AEs) and serious adverse events (SAEs) related to the treatment, including their severity and duration. Adverse events will be classified according to the NIH Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
The Multiple Sclerosis Functional Composite (MSFC) score | From enrollment to the end of treatment at 12 months
  The Multiple Sclerosis Functional Composite (MSFC) is a three-part quantitative objective measure of neurologic function, measuring leg (timed 25-foot walk [25FTW] measured in seconds), arm (nine-hole peg test [9HPT] measured in seconds), and cognitive (three-second paced auditory serial addition test [PASAT3] measured in z-score) functions. The MSFC is a continuous scale that is a composite of the scores of its three parts. A change of 20% or more of the total score (the MSFC composite) or any of its individual component parts (25FTW, 9HPT, PASAT3) is considered clinically significant.
The Six-minute Walk Test | From enrollment to the end of treatment at 12 months
  The maximum distance walked in 6 minutes is measured. If the patient cannot complete the 6-minute walk then the measurement becomes the total time walked. A 20% change in the distance walked in 6 minutes for those who complete the 6-minute walk, or a 20% change in the total time walked for those who cannot, will be considered clinically significant.
The Expanded Disability Status Scale (EDSS) | From enrollment to the end of treatment at 12 months
  The Expanded Disability Status Scale (EDSS) score ranges from 0 to 10.0, with higher scores indicating a greater degree of disability.25 Participants will undergo EDSS assessments at baseline, 6 months, and 12 months. A reduction in EDSS score by 1 point for baseline scores ≤5.5 and by 0.5 points for baseline scores ≤6.0 will indicate a reduction in disability, and vice versa for disability progression.
The Multiple Sclerosis Quality of Life-54 (MSQoL-54) | From enrollment to the end of treatment at 12 months
  The Multiple Sclerosis Quality of Life-54 (MSQoL-54) is a health-related quality of life (HRQoL) questionnaire specifically designed for people with multiple sclerosis (MS). The MSQoL-54 generates 12 subscales and 2 composite scores.
  Scoring:
  1. Item scores range from 1 to 6, depending on the question format.
  2. Raw scores for each subscale are calculated by averaging item responses.
  3. Transformed scores: These raw scores are converted to a 0-100 scale, where 0 represents the worst possible health and 100 represents the best possible health.
  4. Composite scores for physical and mental health are calculated by averaging the relevant subscale scores.
  Interpretation:
  * Higher scores indicate better quality of life.
  * The physical health composite reflects mobility, energy, and physical pain.
  * The mental health composite covers emotional well-being, cognitive function, and social interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdelrazek, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosner M, Horer S, Feichtinger M, Hengstschlager M. Multipotent fetal stem cells in reproductive biology research. Stem Cell Res Ther. 2023 Jun 7;14(1):157. doi: 10.1186/s13287-023-03379-4. PMID 37287077
- [Background] Lassmann H. Pathogenic Mechanisms Associated With Different Clinical Courses of Multiple Sclerosis. Front Immunol. 2019 Jan 10;9:3116. doi: 10.3389/fimmu.2018.03116. eCollection 2018. PMID 30687321